

Optimizing Online Purchasing of Fruits, Vegetables, and Legumes for Low-Income Families

NCT07071753

**Document Date: 01/22/2026** 



## Child Assent Form for IRB-FY2022-6623

(To be read aloud to the child)

Hi! My name is [identify yourself to the child by name]. I work with caregivers and children, and I'm also a student. Right now, I'm trying to learn more about how the foods that kids' caregivers bring home might help kids grow up healthy.

If you agree to be in the study, we will ask to check how tall you are, how much you weigh, and we'll do a quick finger scan to learn more about your body. It won't hurt and only takes a few minutes. You may be helping us understand how what grown-ups bring home to eat can help kids like you stay healthy.

If you agree to help us, your teacher and classmates won't know what we talked about or measured. And if you decide to help us or if you say "no," it won't change anything about school or how anyone treats you.

There are no right or wrong answers. You can talk with your caregivers before you decide. I'll also ask your caregivers if it's okay for you to be in the study, but even if they say "yes," you can still say "no." If you don't want to be in the study, that's totally fine. If you start and later want to stop, that's okay too—no one will be upset.

Also, no one else—not even your caregivers—will know the details of what we measured or talked about.

You can ask me any questions now, or later if you think of something. You can call me, or you can ask your caregivers or teacher to call me at: [insert telephone number].

Would you like to help us today?

[Child answers yes or no; only a definite "yes" may be taken as assent to participate.]